CLINICAL TRIAL: NCT03983525
Title: The Effect of Gojiberry Intake (Lycium Barbarium) on Macular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1220178
Record Dates: First submitted 2019-06-07; First posted 2019-06-12 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Macular Pigment Optical Density
MeSH Terms: interventions — Lutein

STUDY DESIGN:
Intervention Model Description: Randomized paralleled arm clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Goji berry (Experimental): The study will include three study visits over a 90 days period, with study visit one (SV1) occurring at day 0 SV2 conducted at day 45, and SV3 conducted at day 90. The participant will be provided with either a 45-day supply of goji berries and will be asked to consume the given items five days per week. After the 45-day intake period, the participants will return to the lab for SV2 and then be given a new 45-day supply of items to consume until the end of the 90 day test period (SV3).
  Interventions: Dietary Supplement: Goji berry
- Lutein + zeaxanthin supplementation (Active Comparator): The study will include three study visits over a 90 days period, with study visit one (SV1) occurring at day 0. SV2 conducted at day 45, and SV3 conducted at day 90. The participant will be provided with L/Z supplements which contains 6 mg of lutein and 4 mg of zeaxanthin and will be asked to consume the given items five days per week. After the 45-day intake period, the participants will return to the lab for SV2 and then be given a new 45-day supply of items to consume until the end of the 90 day test period (SV3).
  Interventions: Dietary Supplement: Lutein + zeaxanthin supplementation

INTERVENTIONS:
Dietary Supplement: Goji berry — Those who are eligible for enrollment will be required to participate in three study visits over a three-month period, with each visit lasting approximately one and half hour. The three study visits will be separated by 45 +/- 2 days. During each study period, the participants are required to take 28 grams of goji berry once a day, five times per week, and will complete a set of 24 hour dietary recall, using an online automated self-administered recall system known as the ASA24.
  Arms: Goji berry
Dietary Supplement: Lutein + zeaxanthin supplementation — Those who are eligible for enrollment will be required to participate in three study visits over a three-month period, with each visit lasting approximately one and half hour. The three study visits will be separated by 45 +/- 2 days. During each study period, the participants are required to take one capsule of lutein + zeaxanthin supplementation once a day, five times per week, and will complete a set of 24 hour dietary recall, using an online automated self-administered recall system known as the ASA24.
  Arms: Lutein + zeaxanthin supplementation

SUMMARY:
Objective: To evaluate the effects of goji berry intake for three months on macular pigment ocular density (MPOD) between 45 and 65 years old.

Specific Aims:

Determine if goji berry intake for 90 days, 5 times per week, will:

* result in favorable changes in macular pigment optical density (MPOD), as measured using heterochromatic flicker photometry (HFP), in adults aged from 45 to 65 years old.
* impact the carotenoid distribution in the skin.
* will change the fermentation capacity of the gut microbiota.

The investigators hypothesize that the intake of 28 grams of goji berry for 90 days, 5 days per week will significantly increase MPOD after three months, compared to baseline values. In contrast, the investigators hypothesize that a dietary supplement of lutein and zeaxanthin will not alter MPOD.

DETAILED DESCRIPTION:
Prior to enrollment, all volunteers that meet the initial inclusion and exclusion based on a telephone interview will be asked to participate in a clinical screening visit, which will assess the subject's overall health, and whether the individual meets the inclusion and exclusion criteria. To determine normal eye health, subjects will provide a statement from their optometrist verifying normal functioning. The study will be conducted in the Ragle Human Nutrition Research Center on the UC Davis campus. The participants will be consented into the study. For those who are not familiar with goji berry, a sample tasting will be provided. In addition, each volunteer will be asked to complete a diet and health habits questionnaire. The first study visit will begin on the same day after the screening visit is done.

The study will be a randomized, controlled, parallel arm design with two groups: goji berry or lutein/zeaxanthin (L/Z) supplement. Participants will be randomly assigned to one of the two groups using a block design that will place an approximately similar number of males and females in each group. The randomization will be conducted by an online tool called Research Randomizer.

The study will include three study visits over a 90 days period, with study visit one (SV1) occurring at day 0, SV2 conducted at day 45, and SV3 conducted at day 90. The first study visit will occur immediately after consent is completed.

Depending on group assignment, the participant will be provided with either a 45-day supply of goji berries or L/Z supplements which contains 6 mg of lutein and 4 mg of zeaxanthin and will be asked to consume the given items five days per week. After the 45-day intake period, the participants will return to the lab for SV2 and then be given a new 45-day supply of items to consume until the end of the 90 day test period (SV3). Participants will complete a log in order to verify compliance. Dietary recall will be collected by using the Automated Self-Administered 24-hour dietary assessment (ASA24) web-based tool between each SV.

MPOD measurement - MPOD will be assessed by the psychophysical method of HFP technology (Macular Metrics, Providence, RI). Participants will watch a 20 minutes long video of a description of HFP. After adapting to the dark for seven minutes, participants will be asked to rest their head on a chin rest and look at a blue background field for three minutes. Prior to each test, the light intensity from each wavelength will be calibrated with a photodiode. The flicker frequency is selected for each subject based on preliminary tests of flicker sensitivity. The observer's task is to eliminate or minimize the flicker by turning a dial that changes the intensity of the 460-nm light. They will be asked to do this when looking directly at the flickering light and also when looking at a fixation point so that the stimulus can be presented in the periphery.

Skin carotenoid measurement - the carotenoid content in the skin will be measured through a finger-scanning device using reflection spectroscopy (this process does not capture fingerprints) called the Veggie Meter (VM). This noninvasive method of measuring skin carotenoid levels has been validated to reflect plasma carotenoid concentrations.

Breath Hydrogen measurement - the participant will be asked to do one short exhalation (about 2-3 seconds) into a collection tube. Their breath sample will be analyzed for hydrogen and methane that are produced by fermentation of carbohydrates (including fiber) in the digestive tract.

Compliance will be assessed verbally and through self-reported logs indicating consumption of the product. Dietary recall will be collected by using the Automated Self-Administered 24-hour dietary assessment (ASA24) web-based tool during each study arm, and a weekly log book of digestive tract symptoms, which will record a typical symptom such as bloating, gas, intestinal cramps, and loose stools.

ELIGIBILITY:
Inclusion:

Male and female:45-65 years Willing and able to comply with the study protocols Normal macular condition verified by optometry office Stable on prescription medication use, for at least the past 6 months, as approved by the study physician

Exclusion:

Dislike of or allergy to goji berry Self-reported diabetes, renal or liver disease, heart disease, which includes cardiovascular events and stroke, cancer, malabsorption problems, substance abuse or eye diseases

Smoking:

* Current smokers
* Those that have smoked within the past year
* Former smokers with greater than a 20 pack-year history of smoking within the past 20 years Indications of substance or alcohol abuse Current or planned use of blood thinner (eg. Coumadin, Warfarin) at any time during study

Currently taking zeaxanthin or lutein supplements Use of multi-vitamin and mineral supplements other than a general formula that provides up to 100% of the Daily Value Not willing to stop dietary supplement use at least one month prior to study enrollment Currently taking drugs for management of lipids, glucose or blood pressure statin drugs A current enrollee in a clinical research study

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Macular pigment ocular density (MPOD) | 90 days
  MPOD measurement - MPOD will be assessed by the psychophysical method of HFP technology (Macular Metrics, Providence, RI). Participants will watch a 20 minutes long video of a description of HFP. After adapting to the dark for seven minutes, participants will be asked to rest their head on a chin rest and look at a blue background field for three minutes. Prior to each test, the light intensity from each wavelength will be calibrated with a photodiode. The flicker frequency is selected for each subject based on preliminary tests of flicker sensitivity. The observer's task is to eliminate or minimize the flicker by turning a dial that changes the intensity of the 460-nm light. They will be asked to do this when looking directly at the flickering light and also when looking at a fixation point so that the stimulus can be presented in the periphery.

SECONDARY OUTCOMES:
Skin carotenoids concentration | 90 days
  Skin carotenoid measurement - the carotenoid content in the skin will be measured through a finger-scanning device using reflection spectroscopy (this process does not capture fingerprints) called the Veggie Meter (VM). This noninvasive method of measuring skin carotenoid levels has been validated to reflect plasma carotenoid concentrations.
Gut fermentation measured as the hydrogen content in the breath | 90 days
  Breath Hydrogen measurement - the participant will be asked to do one short exhalation (about 2-3 seconds) into a collection tube. Their breath sample will be analyzed for hydrogen and methane that are produced by fermentation of carbohydrates (including fiber) in the digestive tract.

CONTACTS AND LOCATIONS:
Locations (1):
- Regal Human Nutrition Research Center, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No